CLINICAL TRIAL: NCT00173212
Title: Proliferation of Endometrial Stromal Cells in Adenomyosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700522; NTUH.95-000357
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-05

CONDITIONS: Endometriosis
Keywords: adenomyosis; cell proliferation; Immunocytochemistry
MeSH Terms: conditions — Endometriosis; Adenomyosis; Hyperplasia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Adenomyosis refers to the presence of endometrial glands and stroma that is haphazardly deep within the myometrium. However, the etiology and pathologic mechanism responsible for adenomyosis are not yet very well known. Our previous results revealed that the expression of killer inhibitory receptors on natural killer cells was decreased in eutopic endometrium in women with adenomyosis. It implies that the formation of adenomyosis might be due to abnormal endometrial tissues, but not the aberrant local immunological dysfunction in myometrium. Our further investigation revealed that in vitro coculture of macrophages and endometrial stromal cells (ESCs) increase the expression of IL-6 mRNA in ESC, which might further enhance the proliferation of ESC and subsequently result in the formation of ectopic endometrial implants in adenomyosis.

Abnormal cell proliferation has been generally found in the tumorigenesis, including the formation of endometriosis. Adenomyosis is considered to have a similar pathophysiology with endometriosis, and it must be interesting to examine whether there is abnormal cell proliferation in the eutopic endometrium of adenomyosis. Lipopolysaccharide (LPS) was found to promote proliferation of ESCs via induction of TNF-a and IL-8 expression, whereas IFN-g significantly inhibited ESCs proliferation. Therefore, whether abnormal cell proliferation occurs under the effects of LPS and IFN-g in the eutopic endometrium of adenomyosis needs further clarification.

Adenomyosis preferentially affects women between the ages of 35 and 50 years, and the symptoms subside gradually after menopause. It is well known that there is a close conjunction between estrogen and adenomyosis. Estradiol (E2) was demonstrated to induce endometrial cell proliferation, whereas medroxyprogesterone (MPA) inhibited endometrial cell proliferation via antagonizing estrogenic effects. Experiments to investigate these steroid effects on ESC proliferation in vitro in the eutopic endometrium of adenomyosis are of clinical relevance.

In this study, we try to collect endometrial tissues from women with and without adenomyosis, and then purify ESCs from endometrium. ESCs are cultured for 2 days with the supplement of LPS, IFN-gamma, Estradiol, MPA and Estradiol+MPA. Quantification of cell proliferation was done with Cell Proliferation Assay Kit and immunocytochemical detection of Ki-67, in an attempt to examine the cell proliferation of ESCs in women with adenomyosis.

DETAILED DESCRIPTION:
Eutopic endometrium was obtained and separated into single endometrial stromal cell (ESC) in women with adenomyosis (study group) and without adenomyosis (control group).

ESCs are cultured for 2 days with the supplement of LPS, IFN-gamma, Estradiol, MPA and Estradiol+MPA.

Quantification of cell proliferation was done with Cell Proliferation Assay Kit and immunocytochemical detection of Ki-67.

ELIGIBILITY:
Inclusion Criteria:

* women with adenomyosis
* at early- to mid-secretory phases

Exclusion Criteria:

* postmenopausal
* malignancy

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45
Dates: Start 2005-09; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Jehn-Hsiahn Yang, M.D., Principal Investigator — Department of Obstetrics and Gynecology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan